CLINICAL TRIAL: NCT00950599
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 2 Trial to Evaluate the Safety and Efficacy of BMS-477118 as Monotherapy in Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: Study of Multiple Doses of Saxagliptin (BMS-477118)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV181-008
Record Dates: First submitted 2009-07-31; First posted 2009-08-03 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Saxagliptin (2.5 mg) (Experimental)
  Interventions: Drug: Saxagliptin
- Saxagliptin (5 mg) (Experimental)
  Interventions: Drug: Saxagliptin
- Saxagliptin (10 mg) (Experimental)
  Interventions: Drug: Saxagliptin
- Saxagliptin (20 mg) (Experimental)
  Interventions: Drug: Saxagliptin
- Saxagliptin (40 mg) (Experimental)
  Interventions: Drug: Saxagliptin
- Saxagliptin (100 mg) (Experimental)
  Interventions: Drug: Saxagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saxagliptin — Tablets, Oral, 2.5 mg, once daily, 12 weeks
  Other Names: BMS-477118
  Arms: Saxagliptin (2.5 mg)
Drug: Saxagliptin — Tablets, Oral, 5 mg, once daily, 12 weeks
  Other Names: BMS-477118
  Arms: Saxagliptin (5 mg)
Drug: Saxagliptin — Tablets, Oral, 10 mg, once daily, 12 weeks
  Other Names: BMS-477118
  Arms: Saxagliptin (10 mg)
Drug: Saxagliptin — Tablets, Oral, 20 mg, once daily, 12 weeks
  Other Names: BMS-477118
  Arms: Saxagliptin (20 mg)
Drug: Saxagliptin — Tablets, Oral, 40 mg, once daily, 12 weeks
  Other Names: BMS-477118
  Arms: Saxagliptin (40 mg)
Drug: Saxagliptin — Tablets, Oral, 100 mg, once daily, 6 weeks
  Other Names: BMS-477118
  Arms: Saxagliptin (100 mg)
Drug: Placebo — Tablets, Oral, 0 mg, once daily, 6 and 12 weeks
  Arms: Placebo

SUMMARY:
To evaluate the positive efficacy trend among doses of saxagliptin (BMS-477118) in subjects with Type 2 diabetes mellitus by assessing the change from baseline in HbA1c following 12 weeks of double-blind treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes who are drug-naive
* Screening HbA1c ≥ 6.8% and ≤ 9.7%
* Screening fasting or random C-peptide > 0.5 ng/mL
* < 35 years old must be negative for anti-GAD antibodies
* Body Mass Index < 35 kg/m2

Exclusion Criteria:

* Symptoms of poorly controlled diabetes
* History of diabetic ketoacidosis, hyperosmolar nonketotic coma, or insulin therapy within one year of screening
* Receipt of oral antihyperglycemic medications for more than six months in total since diagnosis
* Significant cardiovascular history

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2003-05; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Background] Rosenstock J, Sankoh S, List JF. Glucose-lowering activity of the dipeptidyl peptidase-4 inhibitor saxagliptin in drug-naive patients with type 2 diabetes. Diabetes Obes Metab. 2008 May;10(5):376-86. doi: 10.1111/j.1463-1326.2008.00876.x. Epub 2008 Mar 18. PMID 18355324

RESULTS

PARTICIPANT FLOW:
Groups:
- Saxagliptin 2.5 mg (0-40 mg Cohort): The Saxagliptin 2.5 mg group includes data from subjects randomized to receive blinded Saxagliptin 2.5 mg for 12 weeks
- Saxagliptin 5 mg (0-40 mg Cohort): The Saxagliptin 5 mg group includes data from subjects randomized to receive blinded Saxagliptin 5 mg for 12 weeks.
- Saxagliptin 10 mg (0-40 mg Cohort): The Saxagliptin 10 mg group includes data from subjects randomized to receive blinded Saxagliptin 10 mg for 12 weeks.
- Saxagliptin 20 mg (0-40 mg Cohort): The Saxagliptin 20 mg group includes data from subjects randomized to receive blinded Saxagliptin 20 mg for 12 weeks.
- Saxagliptin 40 mg (0-40 mg Cohort): The Saxagliptin 40 mg group includes data from subjects randomized to receive blinded Saxagliptin 40 mg for 12 weeks.
- Placebo (0-40 mg Cohort): The placebo group includes data from subjects randomized to receive blinded placebo for 12 weeks.
- Saxagliptin 100 mg (0 & 100 mg Cohort): The Saxagliptin 100 mg group includes data from subjects randomized to receive blinded Saxagliptin 100 mg for 6 weeks.
- Placebo (0 & 100 mg Cohort): The placebo group includes data from subjects randomized to receive blinded placebo for 6 weeks.
- Saxa 0-40 mg Cohort (Follow-up Period): The follow-up period is 4 weeks and includes: subjects completing 12 weeks of double-blind dosing (received single blind placebo); subjects who met the hyperglycemic rescue criteria (received open-label metformin in addition to placebo); subjects meeting hyperglycemic discontinuation criteria (received open-label metformin); and subjects who discontinued the double-blind period for reasons other than hyperglycemia (received metformin only if clinically indicated). Open-label metformin was (initiated at 500 mg per day and titrated in 500 mg increments after 2 weeks or as clinically indicated). Additional or alternative antihyperglycemic agents were permitted during the follow-up period as clinically indicated.
- Saxa 0 & 100 mg Cohort (Follow-up Period): The follow-up period is 4 weeks and includes: subjects completing 6 weeks of double-blind dosing (received single blind placebo); subjects who met the hyperglycemic rescue criteria (received open-label metformin in addition to placebo); subjects meeting hyperglycemic discontinuation criteria (received open-label metformin); and subjects who discontinued the double-blind period for reasons other than hyperglycemia (received metformin only if clinically indicated). Open-label metformin was (initiated at 500 mg per day and titrated in 500 mg increments after 2 weeks or as clinically indicated). Additional or alternative antihyperglycemic agents were permitted during the follow-up period as clinically indicated.
Period: Double-Blind Treatment Period
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort) | Saxa 0-40 mg Cohort (Follow-up Period) | Saxa 0 & 100 mg Cohort (Follow-up Period)
Started | 55 | 47 | 63 | 54 | 52 | 67 | 44 | 41 | 0 | 0
Completed | 48 (Completed 12 weeks of treatment) | 37 (Completed 12 weeks of treatment) | 54 (Completed 12 weeks of treatment) | 43 (Completed 12 weeks of treatment) | 45 (Completed 12 weeks of treatment) | 55 (Completed 12 weeks of treatment) | 44 (Completed 12 weeks of treatment) | 35 (Completed 12 weeks of treatment) | 0 | 0
Not Completed | 7 | 10 | 9 | 11 | 7 | 12 | 0 | 6 | 0 | 0
Not completed — Administrative reason by sponsor | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 5 | 5 | 7 | 3 | 6 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0
Not completed — Poor/Noncompliance | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Subject no longer meets study criteria | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Subject Withdrew consent | 4 | 3 | 3 | 1 | 1 | 2 | 0 | 3 | 0 | 0
Period: Follow-Up Period
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort) | Saxa 0-40 mg Cohort (Follow-up Period) | Saxa 0 & 100 mg Cohort (Follow-up Period)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 309 (those completing double blind period (DB) + those rescued/discontinued from DB due to hyperglycemia) | 80 (those completing double blind period (DB) + those rescued/discontinued from DB due to hyperglycemia)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 296 | 78
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Poor/Noncompliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Subject withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort) | Total
Number analyzed (Participants) | 55 | 47 | 63 | 54 | 52 | 67 | 44 | 41 | 423
Age, Customized [Number; unit: participants]
  <65 years | 50 | 39 | 54 | 50 | 41 | 55 | 38 | 35 | 362
  >= 65 years | 5 | 8 | 9 | 4 | 11 | 12 | 6 | 6 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 22 | 23 | 16 | 22 | 25 | 17 | 18 | 176
  Male | 22 | 25 | 40 | 38 | 30 | 42 | 27 | 23 | 247

OUTCOME MEASURES:

1. Primary Outcome: Analysis of Test for Positive Efficacy Trend in Change From Baseline in Hemoglobin A1c (A1C) at Week 12 in the 0-40 mg Cohort
Description: Positive efficacy trend among doses of saxagliptin by assessing the adjusted mean change from baseline in A1C in the 0-40 mg cohort. The unit of measurement for A1C is percent.
Time Frame: Baseline, Week 12
Population: Randomized participants. To be included in analysis of positive efficacy trend in change from baseline to Week 12 Last Observation Carried Forward (LOCF), participants must have had a baseline and at least 1 post-baseline measurement.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobins
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 51 | 42 | 60 | 51 | 50 | 62
percentage of glycosylated hemoglobins | -0.67 (0.80) | -0.95 (0.97) | -0.81 (0.91) | -0.74 (0.93) | -0.78 (1.04) | -0.29 (0.82)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg (0-40 mg Cohort) vs Saxagliptin 5 mg (0-40 mg Cohort) vs Saxagliptin 10 mg (0-40 mg Cohort) vs Saxagliptin 20 mg (0-40 mg Cohort) vs Saxagliptin 40 mg (0-40 mg Cohort) vs Placebo (0-40 mg Cohort); A test for log-linear trend across saxagliptin doses was performed using a linear contrast among the saxagliptin doses from an analysis of covariance (ANCOVA) model. The ANCOVA model was the same model used for the first secondary endpoint; Test type: Superiority or Other; p = 0.9888, Kruskal-Wallis — A significance level of alpha = 0.05 was used for the trend test; ANCOVA Model: post-pre=pre treatment

2. Primary Outcome: Change From Baseline in A1C at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in A1C achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: Randomized participants. To be included in analysis of change from baseline to Week 12 Last Observation Carried Forward (LOCF), participants must have had a baseline and at least 1 post-baseline measurement.
Measure: Mean (Standard Error); unit: percentage of glycosylated hemoglobins
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 51 | 42 | 60 | 51 | 50 | 62
percentage of glycosylated hemoglobins | -0.72 (0.12) | -0.90 (0.14) | -0.81 (0.11) | -0.74 (0.12) | -0.80 (0.12) | -0.27 (0.11)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg (0-40 mg Cohort) vs Saxagliptin 5 mg (0-40 mg Cohort) vs Saxagliptin 10 mg (0-40 mg Cohort) vs Saxagliptin 20 mg (0-40 mg Cohort) vs Saxagliptin 40 mg (0-40 mg Cohort) vs Placebo (0-40 mg Cohort); Test type: Superiority or Other; p = 0.9888, ANCOVA — Positive efficacy trend among doses of saxagliptin by assessing the adjusted mean change from baseline in A1C in the 0-40 mg cohort; ANCOVA Model: post-pre=pretreatment. Contrast Coefficients: -2, -1, 0, 1 2

3. Secondary Outcome: Change From Baseline in A1C at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in A1C achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: Randomized participants. To be included in analysis of change from baseline to Week 6 Last Observation Carried Forward (LOCF), participants must have had a baseline and at least 1 post-baseline measurement.
Measure: Mean (Standard Error); unit: percentage of glycosylated hemoglobins
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 45 | 40 | 54 | 51 | 46 | 57 | 43 | 35
percentage of glycosylated hemoglobins | -0.71 (0.09) | -0.72 (0.10) | -0.67 (0.09) | -0.68 (0.09) | -0.82 (0.09) | -0.33 (0.08) | -1.09 (0.09) | -0.36 (0.09)

4. Secondary Outcome: Change From Baseline in Fasting Serum Glucose (FSG) at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in FSG achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 50 | 46 | 61 | 53 | 50 | 63 | 43 | 37
mg/dL | -10.71 (3.68) | -18.63 (3.82) | -16.10 (3.32) | -14.66 (3.57) | -18.34 (3.67) | -6.20 (3.26) | -26.33 (3.53) | -3.29 (3.81)

5. Secondary Outcome: Change From Baseline in FSG at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in FSG achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 50 | 46 | 61 | 53 | 50 | 63
mg/dL | -10.85 (4.61) | -21.68 (4.80) | -15.91 (4.16) | -13.61 (4.48) | -16.36 (4.60) | 2.81 (4.10)

6. Secondary Outcome: Change From Baseline in Fructosamine at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in fructosamine achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 53 | 44 | 61 | 54 | 49 | 62 | 44 | 36
umol/L | -21.02 (3.91) | -21.87 (4.29) | -24.72 (3.65) | -23.96 (3.88) | -26.03 (4.07) | -9.26 (3.62) | -28.03 (3.74) | -0.16 (4.13)

7. Secondary Outcome: Change From Baseline in Fructosamine at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in fructosamine achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: umol/L
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 54 | 44 | 61 | 54 | 50 | 62
umol/L | -20.89 (4.64) | -25.23 (5.14) | -21.31 (4.36) | -22.30 (4.64) | -26.30 (4.82) | -8.57 (4.33)

8. Secondary Outcome: Change From Baseline in Insulin at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in fasting insulin achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0, 100 mg Cohort) | Placebo (0, 100 mg Cohort)
Number analyzed (Participants) | 45 | 42 | 54 | 48 | 44 | 54 | 39 | 36
uU/mL | 1.88 (1.22) | 1.05 (1.26) | -0.99 (1.11) | -0.17 (1.18) | 0.38 (1.23) | 0.08 (1.11) | -2.03 (1.09) | -0.61 (1.13)

9. Secondary Outcome: Change From Baseline in Insulin at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in insulin achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 42 | 30 | 47 | 37 | 41 | 49
uU/mL | 2.38 (1.63) | 1.02 (1.93) | 1.41 (1.54) | 0.76 (1.74) | 2.29 (1.65) | 1.29 (1.51)

10. Secondary Outcome: Change From Baseline in C-peptide at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in C-peptide achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 45 | 42 | 54 | 48 | 44 | 54 | 39 | 36
ng/mL | -0.15 (0.12) | -0.19 (0.13) | -0.06 (0.11) | -0.02 (0.12) | -0.03 (0.13) | -0.08 (0.11) | -0.52 (0.12) | -0.13 (0.13)

11. Secondary Outcome: Change From Baseline in C-peptide at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in C-peptide achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 42 | 30 | 47 | 37 | 41 | 49
ng/mL | -0.04 (0.14) | -0.13 (0.16) | -0.09 (0.13) | 0.01 (0.14) | -0.02 (0.14) | 0.02 (0.13)

12. Secondary Outcome: Change From Baseline in Postprandial Glucose 0-60 Minute Area Under the Curve (AUC) at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucose 0-60 minute AUC response to a liquid meal tolerance test (MTT) achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts. Area Under the Curve (AUC) here is defined as the area under the plot of the serum concentration of glucose against time after ingesting the meal for the first 60 minutes after the subject drinks the liquid meal.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg*min/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 46 | 37 | 55 | 45 | 44 | 59 | 37 | 32
mg*min/dL | -1226 (318) | -1503 (353) | -1312 (290) | -1246 (320) | -1626 (324) | -461 (280) | -2035 (263) | -664 (283)

13. Secondary Outcome: Change From Baseline in Postprandial Glucose 0-60 Minute AUC at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucose 0-60 minute AUC response to a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort. Area Under the Curve (AUC) is defined as the area under the plot of plasma concentration of drug (not logarithm of the concentration) against time after drug administration. The AUC is of particular use in estimating bioavailability of drugs, and in estimating total clearance of drugs.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg*min/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 39 | 29 | 47 | 38 | 40 | 52
mg*min/dL | -1121 (320) | -1505 (369) | -1730 (289) | -1377 (322) | -1520 (314) | 174 (275)

14. Secondary Outcome: Change From Baseline in Postprandial Insulin 0-60 Minute AUC at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) insulin 0-60 minute AUC response to a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts. Area Under the Curve (AUC) is defined as the area under the plot of plasma concentration of drug (not logarithm of the concentration) against time after drug administration. The AUC is of particular use in estimating bioavailability of drugs, and in estimating total clearance of drugs.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: uU*min/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 44 | 37 | 52 | 46 | 42 | 57 | 35 | 32
uU*min/mL | 234.2 (149.5) | 293.2 (162.3) | 120.0 (136.6) | 165.4 (145.3) | 28.8 (152.4) | 164.6 (130.5) | -296.0 (160.4) | 261.9 (167.7)

15. Secondary Outcome: Change From Baseline in Postprandial Insulin 0-60 Minute AUC at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) insulin 0-60 minute AUC response to a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort. Area Under the Curve (AUC) is defined as the area under the plot of plasma concentration of drug (not logarithm of the concentration) against time after drug administration. The AUC is of particular use in estimating bioavailability of drugs, and in estimating total clearance of drugs.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: uU*min/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 39 | 26 | 46 | 39 | 38 | 51
uU*min/mL | 61.2 (179.9) | 283.4 (218.0) | 114.2 (163.6) | 336.8 (177.7) | 195.6 (180.7) | 30.3 (155.6)

16. Secondary Outcome: Change From Baseline in Postprandial C-peptide 0-60 Minute AUC at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) C-peptide 0-60 minute AUC response to a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts. Area Under the Curve (AUC) is defined as the area under the plot of plasma concentration of drug (not logarithm of the concentration) against time after drug administration. The AUC is of particular use in estimating bioavailability of drugs, and in estimating total clearance of drugs.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ng*min/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 44 | 37 | 52 | 46 | 43 | 57 | 34 | 32
ng*min/mL | 0.2 (9.4) | 7.6 (10.3) | -5.5 (8.7) | 5.4 (9.2) | 0.2 (9.5) | -0.8 (8.3) | -19.7 (9.8) | 0.8 (10.1)

17. Secondary Outcome: Change From Baseline in Postprandial C-peptide 0-60 Minute AUC at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (postprandial) C-peptide 0-60 minute AUC response to a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort. Area Under the Curve (AUC) is defined as the area under the plot of plasma concentration of drug (not logarithm of the concentration) against time after drug administration. The AUC is of particular use in estimating bioavailability of drugs, and in estimating total clearance of drugs.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng*min/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 39 | 26 | 46 | 39 | 38 | 51
ng*min/mL | -8.1 (11.5) | 4.8 (14.0) | -1.6 (10.5) | 7.1 (11.4) | -3.4 (11.6) | -4.0 (10.0)

18. Secondary Outcome: Change From Baseline in 15-minute Postprandial Glucose at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucose 15 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 43 | 35 | 52 | 48 | 40 | 51 | 39 | 34
mg/dL | -15.24 (5.22) | -16.53 (5.75) | -16.78 (4.72) | -14.35 (4.92) | -26.03 (5.38) | -9.30 (4.76) | -25.99 (4.30) | -6.80 (4.61)

19. Secondary Outcome: Change From Baseline in 30-minute Postprandial Glucose at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial glucose 30 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 43 | 34 | 52 | 48 | 42 | 51 | 39 | 33
mg/dL | -23.45 (6.09) | -29.31 (6.80) | -25.32 (5.52) | -23.93 (5.74) | -30.60 (6.12) | -7.81 (5.57) | -36.33 (4.99) | -10.94 (5.42)

20. Secondary Outcome: Change From Baseline in 60-minute Postprandial Glucose at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucose 60 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 43 | 33 | 52 | 48 | 42 | 51 | 38 | 35
mg/dL | -28.45 (6.85) | -39.99 (7.80) | -27.51 (6.21) | -24.32 (6.48) | -34.44 (6.90) | -4.96 (6.29) | -44.58 (5.65) | -17.22 (5.88)

21. Secondary Outcome: Change From Baseline in 15-minute Postprandial Glucose at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucose 15 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 30 | 49 | 38 | 41 | 51
mg/dL | -14.89 (4.78) | -16.45 (5.58) | -19.57 (4.35) | -18.70 (4.94) | -20.75 (4.77) | 0.77 (4.27)

22. Secondary Outcome: Change From Baseline in 30-minute Postprandial Glucose at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial glucose 30 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 30 | 48 | 38 | 42 | 51
mg/dL | -19.79 (5.35) | -24.04 (6.21) | -28.59 (4.92) | -23.56 (5.52) | -20.42 (5.25) | -2.08 (4.76)

23. Secondary Outcome: Change From Baseline in 60-minute Postprandial Glucose at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucose 60 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 30 | 49 | 38 | 41 | 50
mg/dL | -24.42 (6.73) | -35.30 (7.84) | -41.04 (6.14) | -27.54 (6.97) | -33.98 (6.71) | -1.41 (6.08)

24. Secondary Outcome: Change From Baseline in 15-minute Postprandial Insulin at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial insulin 15 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 46 | 38 | 54 | 49 | 45 | 58 | 37 | 33
uU/mL | 5.36 (2.74) | 2.22 (3.02) | 2.47 (2.53) | 3.11 (2.66) | -0.60 (2.77) | 0.60 (2.44) | -1.72 (3.07) | 1.63 (3.25)

25. Secondary Outcome: Change From Baseline in 30-minute Postprandial Insulin at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) insulin 30 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 47 | 37 | 53 | 48 | 47 | 58 | 38 | 33
uU/mL | 5.20 (3.39) | 8.51 (3.81) | 2.04 (3.18) | 1.10 (3.35) | -0.33 (3.40) | 4.82 (3.04) | -4.44 (3.30) | 7.69 (3.54)

26. Secondary Outcome: Change From Baseline in 60-minute Postprandial Insulin at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) insulin 60 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 46 | 37 | 53 | 48 | 44 | 58 | 37 | 34
uU/mL | 2.35 (4.06) | 4.45 (4.49) | 0.25 (3.73) | 4.75 (3.93) | -0.13 (4.11) | 3.33 (3.59) | -8.17 (4.37) | 1.83 (4.56)

27. Secondary Outcome: Change From Baseline in 15-minute Postprandial Insulin at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) insulin 15 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 27 | 48 | 39 | 41 | 54
uU/mL | 2.93 (3.67) | 5.79 (4.49) | 2.87 (3.37) | 6.81 (3.74) | -1.48 (3.65) | 4.70 (3.17)

28. Secondary Outcome: Change From Baseline in 30-minute Postprandial Insulin at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) insulin 30 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 27 | 47 | 39 | 42 | 54
uU/mL | 0.98 (4.09) | 10.71 (5.01) | 2.48 (3.79) | 5.90 (4.16) | 6.14 (4.04) | 1.19 (3.54)

29. Secondary Outcome: Change From Baseline in 60-minute Postprandial Insulin at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) insulin 60 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 27 | 48 | 39 | 39 | 53
uU/mL | 2.62 (4.36) | 4.61 (5.31) | 0.38 (3.95) | 4.99 (4.39) | 2.42 (4.40) | -2.22 (3.80)

30. Secondary Outcome: Change From Baseline in 15-minute Postprandial C-peptide at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) C-peptide 15 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 46 | 38 | 54 | 49 | 45 | 58 | 37 | 33
ng/mL | 0.03 (0.17) | -0.09 (0.19) | -0.12 (0.16) | 0.17 (0.17) | -0.14 (0.17) | -0.13 (0.15) | -0.27 (0.17) | 0.01 (0.18)

31. Secondary Outcome: Change From Baseline in 30-minute Postprandial C-peptide at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) C-peptide 30 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 47 | 37 | 53 | 48 | 47 | 58 | 37 | 33
ng/mL | 0.13 (0.20) | 0.16 (0.23) | -0.01 (0.19) | -0.06 (0.20) | -0.02 (0.21) | 0.03 (0.18) | -0.35 (0.21) | 0.05 (0.22)

32. Secondary Outcome: Change From Baseline in 60-minute Postprandial C-peptide at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) C-peptide 60 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 46 | 37 | 53 | 48 | 45 | 58 | 37 | 34
ng/mL | -0.06 (0.22) | 0.36 (0.25) | -0.16 (0.21) | 0.20 (0.22) | 0.19 (0.22) | 0.24 (0.20) | -0.33 (0.25) | -0.10 (0.26)

33. Secondary Outcome: Change From Baseline in 15-minute Postprandial C-peptide at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) C-peptide 15 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 27 | 48 | 39 | 41 | 54
ng/mL | -0.02 (0.23) | 0.11 (0.28) | -0.12 (0.21) | -0.02 (0.23) | -0.27 (0.23) | 0.07 (0.20)

34. Secondary Outcome: Change From Baseline in 30-minute Postprandial C-peptide at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) C-peptide 30 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 27 | 47 | 39 | 42 | 54
ng/mL | -0.17 (0.23) | 0.27 (0.29) | 0.05 (0.22) | 0.19 (0.24) | 0.12 (0.23) | -0.14 (0.20)

35. Secondary Outcome: Change From Baseline in 60-minute Postprandial C-peptide at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) C-peptide 60 minutes after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 27 | 48 | 39 | 39 | 53
ng/mL | -0.08 (0.26) | 0.18 (0.31) | -0.02 (0.23) | 0.22 (0.26) | 0.01 (0.26) | 0.22 (0.23)

36. Secondary Outcome: Change From Baseline in 15-minute Postprandial Glucose Excursion at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucose excursion (15 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 48 | 39 | 56 | 45 | 44 | 59 | 38 | 33
mg/dL | 1.42 (2.54) | -5.23 (2.82) | -1.15 (2.36) | 3.48 (2.64) | -0.95 (2.65) | -2.37 (2.30) | -1.12 (2.35) | 1.02 (2.52)

37. Secondary Outcome: Change From Baseline in 30-minute Postprandial Glucose Excursion at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucose excursion (30 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 48 | 38 | 55 | 45 | 46 | 59 | 38 | 32
mg/dL | -7.39 (3.24) | -15.91 (3.64) | -6.92 (3.05) | -5.68 (3.34) | -6.89 (3.30) | -2.40 (2.92) | -12.76 (3.87) | -0.79 (4.22)

38. Secondary Outcome: Change From Baseline in 60-minute Postprandial Glucose Excursion at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucose excursion (60 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 48 | 37 | 55 | 45 | 46 | 59 | 38 | 34
mg/dL | -10.08 (4.01) | -23.94 (4.57) | -12.94 (3.75) | -6.10 (4.14) | -11.88 (4.09) | -1.31 (3.63) | -20.69 (4.09) | -8.59 (4.32)

39. Secondary Outcome: Change From Baseline in 15-minute Postprandial Glucose Excursion at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucose excursion (15 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 30 | 48 | 38 | 41 | 53
mg/dL | -1.20 (2.68) | 0.02 (3.13) | 1.63 (2.47) | 3.14 (2.82) | -0.14 (2.68) | 1.89 (2.36)

40. Secondary Outcome: Change From Baseline in 30-minute Postprandial Glucose Excursion at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucose excursion (30 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 30 | 47 | 38 | 42 | 53
mg/dL | -5.99 (3.26) | -5.24 (3.82) | -5.69 (3.06) | -0.73 (3.40) | -0.12 (3.22) | 0.79 (2.87)

41. Secondary Outcome: Change From Baseline in 60-minute Postprandial Glucose Excursion at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucose excursion (60 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 30 | 48 | 38 | 41 | 52
mg/dL | -9.29 (4.26) | -16.51 (5.01) | -19.44 (3.94) | -3.95 (4.43) | -13.83 (4.27) | 0.30 (3.79)

42. Secondary Outcome: Change From Baseline in 15-minute Postprandial Insulin Excursion at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) insulin excursion (15 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 45 | 38 | 53 | 47 | 45 | 57 | 37 | 33
uU/mL | 5.58 (2.53) | -1.04 (2.75) | 2.85 (2.32) | 1.18 (2.47) | 0.11 (2.52) | -0.28 (2.24) | 2.19 (2.62) | 2.67 (2.78)

43. Secondary Outcome: Change From Baseline in 30-minute Postprandial Insulin Excursion at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) insulin excursion (30 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 46 | 37 | 52 | 46 | 47 | 57 | 38 | 33
uU/mL | 4.95 (3.25) | 5.07 (3.61) | 2.40 (3.05) | -0.89 (3.24) | 0.13 (3.23) | 3.23 (2.91) | 0.22 (3.05) | 9.87 (3.27)

44. Secondary Outcome: Change From Baseline in 60-minute Postprandial Insulin Excursion at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) insulin excursion (60 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 45 | 37 | 52 | 46 | 44 | 57 | 37 | 34
uU/mL | 4.03 (3.93) | 1.84 (4.29) | 0.75 (3.60) | 2.28 (3.83) | -0.16 (3.93) | 1.82 (3.47) | -3.61 (3.78) | 4.19 (3.95)

45. Secondary Outcome: Change From Baseline in 15-minute Postprandial Insulin Excursion at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) insulin excursion (15 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 27 | 47 | 39 | 41 | 52
uU/mL | 2.33 (3.08) | 5.26 (3.76) | 1.98 (2.85) | 3.56 (3.14) | -1.49 (3.05) | 4.42 (2.71)

46. Secondary Outcome: Change From Baseline in 30-minute Postprandial Insulin Excursion at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) insulin excursion (30 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 27 | 46 | 39 | 42 | 52
uU/mL | -0.23 (3.47) | 10.17 (4.25) | 1.43 (3.25) | 3.35 (3.53) | 5.36 (3.44) | -0.70 (3.06)

47. Secondary Outcome: Change From Baseline in 60-minute Postprandial Insulin Excursion at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) insulin excursion (60 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 27 | 47 | 39 | 39 | 51
uU/mL | 2.71 (3.97) | 4.85 (4.82) | -0.83 (3.63) | 2.02 (3.99) | 1.44 (4.01) | -3.52 (3.51)

48. Secondary Outcome: Change From Baseline in 15-minute Postprandial C-peptide Excursion at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) C-peptide excursion (15 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 45 | 38 | 53 | 47 | 45 | 57 | 37 | 33
ng/mL | 0.29 (0.14) | -0.08 (0.16) | 0.10 (0.13) | 0.08 (0.14) | 0.01 (0.14) | 0.01 (0.13) | 0.01 (0.15) | 0.17 (0.16)

49. Secondary Outcome: Change From Baseline in 30-minute Postprandial C-peptide Excursion at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) C-peptide excursion (30 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 46 | 37 | 52 | 46 | 47 | 57 | 37 | 33
ng/mL | 0.35 (0.18) | 0.11 (0.20) | 0.23 (0.17) | -0.07 (0.18) | 0.12 (0.18) | 0.09 (0.16) | -0.00 (0.20) | 0.31 (0.21)

50. Secondary Outcome: Change From Baseline in 60-minute Postprandial C-peptide Excursion at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) C-peptide excursion (60 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 45 | 37 | 52 | 46 | 45 | 57 | 37 | 34
ng/mL | 0.27 (0.20) | 0.35 (0.22) | 0.17 (0.19) | 0.12 (0.20) | 0.36 (0.20) | 0.17 (0.18) | 0.04 (0.21) | 0.20 (0.21)

51. Secondary Outcome: Change From Baseline in 15-minute Postprandial C-peptide Excursion at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) C-peptide excursion (15 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 27 | 47 | 39 | 41 | 52
ng/mL | 0.23 (0.16) | 0.42 (0.20) | 0.02 (0.15) | 0.02 (0.17) | -0.04 (0.16) | 0.21 (0.15)

52. Secondary Outcome: Change From Baseline in 30-minute Postprandial C-peptide Excursion at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) C-peptide excursion (30 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 27 | 46 | 39 | 42 | 52
ng/mL | 0.05 (0.20) | 0.58 (0.24) | 0.16 (0.18) | 0.28 (0.20) | 0.32 (0.19) | -0.08 (0.17)

53. Secondary Outcome: Change From Baseline in 60-minute Postprandial C-peptide Excursion at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) C-peptide excursion (60 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin versus placebo at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 41 | 27 | 47 | 39 | 39 | 51
ng/mL | 0.29 (0.22) | 0.59 (0.27) | 0.16 (0.20) | 0.27 (0.22) | 0.20 (0.22) | 0.13 (0.20)

54. Secondary Outcome: Change From Baseline in 30-minute Postprandial Glucagon at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucagon 30 minutes after a MTT achieved at each dose of saxagliptin at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 43 | 30 | 46 | 35 | 41 | 50 | 31 | 30
pg/mL | -11.84 (4.11) | -10.92 (4.93) | -11.26 (3.99) | -5.81 (4.56) | -9.04 (4.21) | -1.98 (3.82) | -14.97 (3.69) | 1.17 (3.75)

55. Secondary Outcome: Change From Baseline in 30-minute Postprandial Glucagon at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucagon 30 minutes after a MTT achieved at each dose of saxagliptin at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 40 | 22 | 37 | 30 | 35 | 43
pg/mL | -8.39 (4.12) | -6.06 (5.57) | -12.64 (4.30) | -17.21 (4.76) | -11.90 (4.41) | -3.64 (3.98)

56. Secondary Outcome: Change From Baseline in 30-minute Postprandial Free Fatty Acids (FFA) at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) FFA 30 minutes after a MTT achieved at each dose of saxagliptin at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mEg/L
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 37 | 35 | 48 | 40 | 39 | 44 | 39 | 32
mEg/L | 0.01 (0.03) | -0.03 (0.03) | -0.07 (0.02) | -0.08 (0.03) | -0.05 (0.03) | -0.02 (0.02) | -0.17 (0.02) | -0.16 (0.02)

57. Secondary Outcome: Change From Baseline in 30-minute Postprandial FFA at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) FFA 30 minutes after a MTT achieved at each dose of saxagliptin at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mEg/L
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 32 | 26 | 44 | 32 | 37 | 41
mEg/L | 0.01 (0.03) | -0.00 (0.03) | -0.06 (0.03) | -0.05 (0.03) | -0.04 (0.03) | -0.00 (0.03)

58. Secondary Outcome: Change From Baseline in 30-minute Postprandial Glucagon Excursion at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucagon excursion (30 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 43 | 29 | 44 | 35 | 40 | 48 | 31 | 28
pg/mL | -5.94 (3.64) | -5.75 (4.42) | -10.39 (3.60) | -3.94 (4.02) | -6.99 (3.76) | 3.58 (3.45) | -8.54 (3.87) | 0.52 (4.07)

59. Secondary Outcome: Change From Baseline in 30-minute Postprandial Glucagon Excursion at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) glucagon excursion (30 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 39 | 21 | 36 | 30 | 35 | 42
pg/mL | -5.96 (3.29) | -4.46 (4.47) | -6.80 (3.42) | -10.36 (3.74) | -8.56 (3.47) | 4.53 (3.17)

60. Secondary Outcome: Change From Baseline in 30-minute Postprandial FFA Excursion at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Adjusted mean change from baseline in postprandial (after mealtime) FFA excursion (30 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mEq/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 34 | 30 | 40 | 34 | 36 | 41 | 39 | 31
mEq/mL | -0.02 (0.02) | 0.01 (0.02) | -0.02 (0.02) | 0.00 (0.02) | 0.02 (0.02) | -0.01 (0.02) | -0.07 (0.02) | -0.12 (0.03)

61. Secondary Outcome: Change From Baseline in 30-minute Postprandial FFA Excursion at Week 12 in the 0-40 mg Cohort
Description: Adjusted mean change from baseline in postprandial (after mealtime) FFA excursion (30 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin at Week 12 in the 0-40 mg cohort.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mEq/mL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 32 | 21 | 40 | 28 | 32 | 38
mEq/mL | -0.01 (0.02) | -0.04 (0.03) | 0.02 (0.02) | -0.01 (0.02) | 0.03 (0.02) | -0.04 (0.02)

62. Secondary Outcome: Change From Baseline in 15-minute Insulinogenic Index at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Mean change from baseline in 15-minute insulinogenic index of a MTT achieved at each dose of saxagliptin at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts. The insulinogenic index is a unitless scale which is a measure of insulin production normalized for the glucose stimulus. Higher numbers mean more beta cell function (improvement). The low value is zero. The highest value obtainable is unknown.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 34 | 20 | 41 | 27 | 31 | 40 | 31 | 23
units on a scale | 0.38 (2.04) | -0.31 (2.41) | 0.45 (1.88) | -0.22 (1.22) | 0.04 (2.00) | 0.22 (1.80) | -0.25 (4.52) | -0.63 (2.77)

63. Secondary Outcome: Change From Baseline in 15-minute Insulinogenic Index at Week 12 in the 0-40 mg Cohort
Description: Mean change from baseline in 15-minute insulinogenic index of a MTT achieved at each dose of saxagliptin at Week 12 in the 0-40 mg cohort. The insulinogenic index is a unitless scale which is a measure of insulin production normalized for the glucose stimulus. Higher numbers mean more beta cell function (improvement). The low value is zero. The highest value obtainable is unknown.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 28 | 16 | 35 | 26 | 26 | 39
units on a scale | 0.50 (2.03) | -0.19 (1.77) | -0.13 (1.91) | -0.34 (1.21) | 0.22 (1.54) | -0.05 (1.38)

64. Secondary Outcome: Change From Baseline in 30-minute Insulinogenic Index at Week 6 in the 0-40 and 0 & 100 mg Cohorts.
Description: Mean change from baseline in 30-minute insulinogenic index of a MTT achieved at each dose of saxagliptin at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts. The insulinogenic index is a unitless scale which is a measure of insulin production normalized for the glucose stimulus. Higher numbers mean more beta cell function (improvement). The low value is zero. The highest value obtainable is unknown.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 34 | 20 | 41 | 27 | 31 | 40 | 31 | 23
units on a scale | 0.44 (1.06) | 0.37 (0.76) | 0.31 (0.77) | 0.18 (0.81) | 0.71 (3.71) | 0.04 (0.72) | 0.46 (1.17) | -0.05 (0.83)

65. Secondary Outcome: Change From Baseline in 30-minute Insulinogenic Index at Week 12 in the 0-40 mg Cohort
Description: Mean change from baseline in 30-minute insulinogenic index of a MTT achieved at each dose of saxagliptin at Week 12 in the 0-40 mg cohort. The insulinogenic index is a unitless scale which is a measure of insulin production normalized for the glucose stimulus. Higher numbers mean more beta cell function (improvement). The low value is zero. The highest value obtainable is unknown.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 28 | 16 | 35 | 26 | 26 | 39
units on a scale | 0.15 (0.99) | 0.84 (2.31) | 0.35 (0.97) | -0.05 (0.50) | 0.25 (0.58) | 0.11 (0.44)

66. Secondary Outcome: Change From Baseline in Matsuda Index at Week 6 in the 0-40 and 0 & 100 mg Cohorts
Description: Mean change from baseline in Matsuda index achieved at each dose of saxagliptin at Week 6 in the 0-40 mg and the 0 & 100 mg cohorts. The Matsuda index is a scale designed to give numbers between 0 and 12, with a linear relationship to other indices of insulin sensitivity. The higher the number, the better the insulin sensitivity (improvement).
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 44 | 36 | 52 | 45 | 42 | 57 | 35 | 31
units on a scale | -0.36 (1.36) | 0.31 (1.27) | -0.04 (2.84) | 0.31 (1.76) | -0.06 (2.49) | -0.25 (1.91) | 0.86 (2.86) | 0.35 (2.45)

67. Secondary Outcome: Change From Baseline in Matsuda Index at Week 12 in the 0-40 mg Cohort
Description: Mean change from baseline in Matsuda index achieved at each dose of saxagliptin at Week 12 in the 0-40 mg cohort. The Matsuda index is a scale designed to give numbers between 0 and 12, with a linear relationship to other indices of insulin sensitivity. The higher the number, the better the insulin sensitivity (improvement).
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 40 | 26 | 45 | 40 | 39 | 51
units on a scale | -0.48 (2.81) | 0.34 (1.21) | 0.27 (3.90) | 0.78 (3.24) | 0.17 (3.68) | -0.15 (1.66)

68. Secondary Outcome: Change From Baseline in A1C at 2 Weeks After Discontinuation of Double-Blind Study Medication in the 0-40 and 0 & 100 mg Cohorts
Description: Mean change from baseline in A1C achieved at each dose of saxagliptin during the Follow-Up period at Week 14 in the 0-40 mg cohort and at Week 8 in the 0 & 100 mg cohort.
Time Frame: Baseline, Week 14
Population: Randomized participants. To be included in analysis of change from baseline to Week 14 (0-40 mg cohort) or Week 8 (0&100 mg cohort), participants must have had a baseline and at least 1 follow-up period measurement. Week 14 and Week 8 assessments are the assessments closest to the respective target dates (or later assessments in the case of a tie).
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobins
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 47 | 39 | 55 | 47 | 46 | 59 | 41 | 32
percentage of glycated hemoglobins | -0.55 (0.93) | -0.84 (1.04) | -0.78 (0.98) | -0.66 (1.03) | -0.69 (1.04) | -0.25 (0.83) | -1.15 (0.76) | -0.45 (0.65)

69. Secondary Outcome: Change From Baseline in A1C at 4 Weeks After Discontinuation of Double-Blind Study Medication in the 0-40 and 0 & 100 mg Cohorts
Description: Mean change from baseline in A1C achieved at each dose of saxagliptin during the Follow-Up period at Week 16 in the 0-40 mg cohort and at Week 10 in the 0 & 100 mg cohort.
Time Frame: Baseline, Week 10, Week 16
Population: Randomized participants. To be included in analysis of change from baseline to Week 16 (0-40 mg cohort) and Week 10 (0&100 mg cohort), participants must have had a baseline and at least 1 follow-up period measurement. Week 16 and Week 10 assessments are the assessments closest to the respective target date (or later assessment in the case of a tie)
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobins
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 47 | 40 | 56 | 42 | 45 | 56 | 41 | 32
percentage of glycated hemoglobins | -0.34 (0.98) | -0.72 (0.96) | -0.64 (0.99) | -0.57 (0.94) | -0.53 (0.97) | -0.24 (0.87) | -1.01 (0.70) | -0.43 (0.80)

70. Secondary Outcome: Change From Baseline in FSG at 2 Weeks After Discontinuation of Double-Blind Study Medication in the 0-40 and 0 & 100 mg Cohorts
Description: Mean change from baseline in FSG achieved at each dose of saxagliptin during Follow-Up period at Week 14 in the 0-40 mg cohort and at Week 8 in the 0 & 100 mg cohort.
Time Frame: Baseline, Week 8, Week 14
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 46 | 39 | 55 | 47 | 47 | 56 | 43 | 32
mg/dL | -1.93 (36.86) | -14.03 (34.62) | -7.58 (29.35) | -11.17 (33.97) | -6.02 (38.40) | -0.75 (29.11) | -14.14 (26.14) | -3.47 (26.80)

71. Secondary Outcome: Change From Baseline in FSG at 4 Weeks After Discontinuation of Double-Blind Study Medication in the 0-40 and 0 & 100 mg Cohorts
Description: Mean change from baseline in FSG achieved at each dose of saxagliptin during the follow-up period at Week 16 in the 0-40 mg cohort and at Week 10 in the 0 & 100 mg cohort.
Time Frame: Baseline, Week 10, Week 16
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 45 | 40 | 54 | 44 | 44 | 55 | 39 | 32
mg/dL | -5.82 (31.60) | -11.55 (33.73) | -6.65 (46.36) | -9.05 (28.62) | -0.91 (33.94) | -2.04 (40.19) | -7.82 (23.88) | -5.97 (21.76)

72. Secondary Outcome: Change From Baseline in Fructosamine at 2 Weeks After Discontinuation of Double-Blind Study Medication in the 0-40 and 0 & 100 mg Cohorts
Description: Mean change from baseline in fructosamine achieved at each dose of saxagliptin during the Follow-up period at Week 14 in the 0-40 mg cohort and at Week 8 in the 0 & 100 mg cohort.
Time Frame: Baseline, Week 8, Week 14
Population: Randomized participants. To be included in analysis of change from baseline to Week 14 or Week 8, participants must have had a baseline and at least 1 post-baseline measurement. The Week 14 and Week 8 assessments are the assessments closest to the respective target dates (or later assessments in the case of a tie).
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 47 | 40 | 56 | 48 | 47 | 58 | 44 | 32
umol/L | -12.40 (35.18) | -19.78 (33.80) | -12.77 (37.92) | -17.10 (39.36) | -12.81 (32.41) | -7.48 (34.15) | -21.86 (31.39) | -5.97 (23.67)

73. Secondary Outcome: Change From Baseline in Fructosamine at 4 Weeks After Discontinuation of Double-Blind Study Medication in the 0-40 and 0 & 100 mg Cohorts
Description: Mean change from baseline in fructosamine achieved at each dose of saxagliptin during the Follow-up period at Week 16 in the 0-40 mg cohort and at Week 10 in the 0 & 100 mg cohort.
Time Frame: Baseline, Week 10, Week 16
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 47 | 41 | 55 | 45 | 44 | 56 | 40 | 32
umol/L | -8.60 (39.61) | -8.02 (37.54) | -11.02 (40.73) | -19.44 (37.39) | -10.14 (31.45) | -7.05 (35.13) | -15.25 (30.78) | -10.00 (24.26)

74. Secondary Outcome: Change From Baseline in A1C at Week 6 by Baseline A1C Category in the 0 & 100 Cohort
Description: Adjusted mean change from baseline in A1C achieved at each dose of saxagliptin at Week 6 in subjects with baseline A1C <7%, ≥7% to <8%, ≥8% to <9%, and ≥9% in the 0 & 100 mg cohort.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 43 | 35
percent
  <7% (n=8; n=12) | -0.61 (0.26) | -0.18 (0.27)
  ≥7% to <8% (n=20; n=8) | -1.01 (0.41) | -0.30 (0.15)
  ≥8% to <9% (n=9; n=11) | -1.14 (0.53) | -0.34 (0.95)
  ≥9% (n=6; n=4) | -2.10 (0.88) | -0.83 (0.31)

75. Secondary Outcome: Change From Baseline in FSG at Week 6 in Subjects by Baseline FSG Category in the 0 & 100 mg Cohort.
Description: Adjusted mean change from baseline in FSG achieved at each dose of saxagliptin at Week 6 in subjects with baseline FSG <140 mg/dL, ≥140 mg/dL to <180 mg/dL, and ≥ 180 mg/dL in the 0 & 100 mg cohort.
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 43 | 37
mg/dL
  < 140 mg/dL (n=17; n=17) | -11.12 (12.51) | 1.29 (12.95)
  140 - < 180 mg/dL (n=17; n=14) | -27.00 (19.47) | 0.07 (26.78)
  ≥180 mg/dL (n=9; n=6) | -56.89 (25.21) | -19.50 (48.14)

76. Secondary Outcome: Change From Baseline in 60 Minute Postprandial Glucose at Week 6 by Baseline Category in the 0 & 100 mg Cohort
Description: Adjusted mean change from baseline in 60-minute postprandial glucose achieved at each dose of saxagliptin at Week 6 in subjects with baseline 60-minute postprandial glucose <140 mg/dL, ≥140 to <200 mg/dL, and ≥200 mg/dL in the 0 & 100 mg cohort.
Time Frame: Baseline, Week 6
Population: Randomized participants. To be included in analysis of change from baseline to Week 6, participants must have had a baseline and at least 1 post-baseline measurement.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 38 | 35
mg/dL
  <140 mg/dL (n=1; n=3) | -18.00 (0.00) | 11.33 (12.10)
  ≥140 to <200 mg/dL (n=17; n=12) | -24.29 (21.44) | -19.25 (25.30)
  ≥200 mg/dL (n=20; n=20) | -62.10 (34.83) | -21.35 (57.10)

77. Secondary Outcome: Percentage of Participants Achieving A1C < 7% at Week 6 in the 0 & 100 mg Cohort
Description: Percentage of participants achieving A1C < 7%, the American Diabetic Association's defined goal for glycemia, at each dose of saxagliptin at Week 6 in the 0 & 100 mg cohort.
Time Frame: Week 6
Population: Randomized participants. To be included in the Week 6 LOCF analysis, subjects must have had at least 1 post-baseline measurement.
Measure: Number; unit: Percentage of Participants
Arm/Group | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 44 | 41
Percentage of Participants | 72 | 49

78. Secondary Outcome: Change From Baseline in 60-minute Postprandial FFA Excursion at Week 6 in the 0 & 100 mg Cohort
Description: Adjusted mean change from baseline in postprandial FFA excursion (60 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin at Week 6 in the 0 & 100 mg cohort. (Note: this analysis was not performed.)
Time Frame: Baseline, Week 6
Population: as for outcome 3
Arm/Group | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 0 | 0

79. Secondary Outcome: Change From Baseline in 60-minute Postprandial Glucagon Excursion at Week 6 in the 0 & 100 mg Cohort
Description: Adjusted mean change from baseline in postprandial glucagon excursion (60 minutes minus 0 minutes) after a MTT achieved at each dose of saxagliptin at Week 6 in the 0 & 100 mg cohort. (Note: this analysis was not performed.)
Time Frame: Baseline, Week 6
Arm/Group | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 0 | 0

80. Secondary Outcome: Discontinuations During the Double-Blind Phase Due to Lack of Glycemic Control
Description: Number of participants discontinuing from the double-blind phase due to lack of glycemic control at Week 4 and Week 6. (Note: this analysis was not performed.)
Time Frame: Week 4, Week 6
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

81. Secondary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths and Discontinuations During the Double-Blind Treatment Period in the 0-40 mg Cohort
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. Related AE=relationship of certain, probable, possible, or missing. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in the development of drug dependency or drug abuse, is an important medical event.
Time Frame: up to Week 12 for AEs; up to 30 days post-double-blind period but prior to follow-up period if any for SAEs and up to 30 days post-double-blind period for Discontinuations
Population: All participants randomized and treated during the double-blind period.
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 55 | 47 | 63 | 54 | 52 | 67
Percentage of participants
  At least one AE | 80.0 | 76.6 | 77.8 | 87.0 | 75.0 | 79.1
  At least one SAE | 1.8 | 0 | 1.6 | 1.9 | 0 | 1.5
  At least one related AE | 14.5 | 23.4 | 22.2 | 25.9 | 23.1 | 23.9
  Deaths | 0 | 0 | 0 | 0 | 0 | 0
  Discontinuations due to AEs | 0 | 2.1 | 1.6 | 1.9 | 3.8 | 1.5

82. Secondary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths and Discontinuations During the Double-Blind Treatment Period in the 0 & 100 mg Cohort
Description: as for outcome 81
Time Frame: up to Week 6 for AEs; up to 30 days post-double-blind period but prior to follow-up period if any for SAEs and up to 30 days post-double-blind period for Discontinuations
Population: All participants randomized and treated during the double-blind period.
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 Cohort)
Number analyzed (Participants) | 44 | 41
Percentage of participants
  At least one AE | 65.9 | 58.5
  At least one SAE | 0 | 0
  At least one related AE | 22.7 | 12.2
  Deaths | 0 | 0
  Discontinuations due to AEs | 0 | 0

83. Secondary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths and Discontinuations During the Follow-up Period in the 0-40 mg Cohort
Description: as for outcome 81
Time Frame: From Week 12 to Week 16 for AEs; up to 30 days post follow-up in both cohorts for SAEs and Discontinuations
Population: All participants treated during the follow-up period.
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Placebo (0-40 mg Cohort)
Number analyzed (Participants) | 50 | 42 | 58 | 48 | 47 | 60
Percentage of participants
  At least one AE | 34.0 | 42.9 | 37.9 | 37.5 | 42.6 | 26.7
  At least one SAE | 0 | 0 | 0 | 2.1 | 0 | 1.7
  At least one related AE | 4.0 | 7.1 | 3.4 | 12.5 | 4.3 | 6.7
  Deaths | 0 | 0 | 0 | 0 | 0 | 0
  Discontinuations due to AEs | 0 | 0 | 0 | 0 | 0 | 0

84. Secondary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths and Discontinuations During the Follow-up Period in the 0 & 100 mg Cohort
Description: as for outcome 81
Time Frame: From Week 6 to Week 10 for AEs; up to 30 days post follow-up in both cohorts for SAEs and Discontinuations
Population: All participants treated during the follow-up period.
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 100 mg (0 & 100 mg Cohort) | Placebo (0 & 100 mg Cohort)
Number analyzed (Participants) | 44 | 36
Percentage of participants
  At least one AE | 31.8 | 33.3
  At least one SAE | 0 | 0
  At least one related SAE | 2.3 | 0
  Deaths | 0 | 0
  Discontinuations due to AEs | 0 | 0

ADVERSE EVENTS:
Arm/Group | Saxagliptin 10 mg (0-40 mg Cohort) | Saxagliptin 100 mg (0 & 100 mg Cohort) | Saxagliptin 2.5 mg (0-40 mg Cohort) | Saxagliptin 20 mg (0-40 mg Cohort) | Saxagliptin 40 mg (0-40 mg Cohort) | Saxagliptin 5 mg (0-40 mg Cohort) | Placebo (0 & 100 mg Cohort) | Placebo (0-40 mg Cohort)
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/44 | 1/55 | 2/54 | 0/52 | 0/47 | 0/41 | 2/67
Other Adverse Events (participants affected / at risk) | 36/63 | 16/44 | 35/55 | 33/54 | 27/52 | 23/47 | 17/41 | 38/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin 10 mg (0-40 mg Cohort) (N=63) | Saxagliptin 100 mg (0 & 100 mg Cohort) (N=44) | Saxagliptin 2.5 mg (0-40 mg Cohort) (N=55) | Saxagliptin 20 mg (0-40 mg Cohort) (N=54) | Saxagliptin 40 mg (0-40 mg Cohort) (N=52) | Saxagliptin 5 mg (0-40 mg Cohort) (N=47) | Placebo (0 & 100 mg Cohort) (N=41) | Placebo (0-40 mg Cohort) (N=67)
Rectocele (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystocele (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin 10 mg (0-40 mg Cohort) (N=63) | Saxagliptin 100 mg (0 & 100 mg Cohort) (N=44) | Saxagliptin 2.5 mg (0-40 mg Cohort) (N=55) | Saxagliptin 20 mg (0-40 mg Cohort) (N=54) | Saxagliptin 40 mg (0-40 mg Cohort) (N=52) | Saxagliptin 5 mg (0-40 mg Cohort) (N=47) | Placebo (0 & 100 mg Cohort) (N=41) | Placebo (0-40 mg Cohort) (N=67)
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 1 | 2 | 2 | 3 | 0 | 1
Hot Flush (Vascular disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 10 | 5 | 8 | 6 | 5 | 4 | 2 | 6
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 5 | 2 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 3 | 0 | 1 | 3 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 4 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 3 | 3 | 3 | 0 | 2 | 2
Influenza (Infections and infestations) | 2 | 0 | 3 | 1 | 2 | 0 | 1 | 3
Sinusitis (Infections and infestations) | 4 | 2 | 2 | 1 | 1 | 2 | 2 | 4
Bronchitis (Infections and infestations) | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 4
Nasopharyngitis (Infections and infestations) | 5 | 1 | 0 | 3 | 6 | 2 | 1 | 5
Urinary Tract Infection (Infections and infestations) | 4 | 4 | 6 | 5 | 2 | 2 | 2 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 0 | 6 | 6 | 0 | 3 | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 1 | 2 | 1 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 4 | 1 | 2 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 6 | 5 | 2 | 3 | 1 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 2 | 3 | 2 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 3 | 3 | 3 | 0 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0 | 1 | 3 | 1 | 2
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 2 | 3 | 0 | 4
Fatigue (General disorders) | 1 | 3 | 2 | 2 | 3 | 0 | 2 | 0
Oedema Peripheral (General disorders) | 4 | 2 | 0 | 1 | 2 | 1 | 1 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.